CLINICAL TRIAL: NCT04501874
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Study to Evaluate the Safety and Efficacy of EMB 001 in Subjects With Moderate-to-Severe Cocaine Use Disorder
Brief Title: A Study to Evaluate EMB 001 in Subjects With Cocaine Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERL-003; 5U01DA038879-03 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cocaine Use Disorder
Keywords: cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EMB-001 Active (Active Comparator): EMB-001 Combination product of 720 mg metyrapone/24 mg oxazepam mg by mouth twice per day for 12 weeks followed by a 1 week taper
  Interventions: Drug: EMB-001
- EMB-001 Placebo (Placebo Comparator): EMB-001 Placebo by mouth twice per day for 12 weeks followed by a 1 week taper
  Interventions: Drug: EMB-001 Placebo

INTERVENTIONS:
Drug: EMB-001 — 720 mg metyrapone/24 mg oxazepam mg BID
  Arms: EMB-001 Active
Drug: EMB-001 Placebo — Inactive comparator
  Arms: EMB-001 Placebo

SUMMARY:
EMB-001 is a combination of 2 drugs: the cortisol synthesis inhibitor, metyrapone (Metopirone®), and the benzodiazepine receptor agonist, oxazepam (original trade name Serax®; now marketed as oxazepam (generic) only).

This is a Phase 2 study in approximately 80 adult subjects with moderate-to-severe Cocaine Use Disorder (CUD).

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, study to compare the safety and efficacy of EMB-001 with a placebo control in approximately 80 subjects with moderate-to-severe CUD. Subjects will receive investigational medicinal product (IMP) during a 12-week, double-blind Treatment Period (Week 2 through Week 13) and a 1-week, double-blind Taper Period (Week 14).

After undergoing study procedures during the Screening and Baseline Periods, subjects who meet inclusion and exclusion criteria will then be randomized in a 1:1 ratio (n=40/arm) to one of the following for the Treatment Period (weeks 2 - 13) on Study Day 8:

* EMB-001 720 mg metyrapone/24 mg oxazepam mg BID, for a total daily dose of 1440 mg metyrapone and 48 mg oxazepam (Active Group)
* Placebo BID, (Placebo Group)

During the Taper Period (week 14), subjects in the Active Group will receive EMB-001 240/8 mg BID; and the Placebo Group will continue to receive placebo. Both groups will change from taking three capsules BID (twice daily) to one capsule BID (twice daily).

There will be a follow-up visit for safety assessments at Week 18.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written informed consent prior to any study procedures
* 18 to 65 years of age
* DSM-5 diagnosis of moderate-to-severe CUD
* Seeking treatment for CUD. Subjects with past rehabilitation attempts are eligible if the most recent rehabilitation attempt ended at least 30 days prior to Screening
* Female subjects must be of non-childbearing potential
* Male subjects must agree to use accepted contraceptive regimens during the study and for at least 90 days after the last dose of the study drug

Key Exclusion Criteria:

* Any significant current medical conditions
* Known hypersensitivity to or intolerance of oxazepam, metyrapone, or any benzodiazepine, or severe hypersensitivity reaction (e.g., angioedema) to any drug
* Heightened likelihood of having adrenal insufficiency in the investigator's or designees' opinion
* Current court-mandated treatment requirement for a substance-use disorder
* Current DSM-5 moderate-to-severe substance use disorder, other than CUD, tobacco or caffeine
* Current DSM-5 opioid or benzodiazepine use disorder of any severity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects must be of non-childbearing potential.
Enrollment: 82 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Continuous Abstinence from Cocaine Use | Week 11 to Week 13
  The Primary Endpoint is the Proportion of Subjects That Successfully Achieve Abstinence From Cocaine During the Last Three Weeks of Treatment using the Timeline Follow Back; days of abstinence, confirmed by Urine benzoylecgonine (BE)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 13 weeks
  Adverse event data (including clinically significant changes in laboratory values) will be compiled for EMB-001 and placebo cohorts.
Reduction in cocaine-use days | Week 2 to Week 13
  Self-report weekly cocaine non-use days by Timeline Follow-Back
Urine confirmation of cocaine use | Week 2 to Week 13
  Qualitative urine BE levels twice per week
Reduction in total Cocaine Craving Questionnaire-Brief score | Week 2 to Week 13
  The Cocaine Craving Questionnaire-Brief (CCQ-B) assesses current cocaine craving in routine clinical practice. The CCQ-B is a 10 item questionnaire and items are scored on a one to seven scale. Total responses are then divided by 10 to achieve a total craving score between 1.0 (least craving) to 7.0 (most craving).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce McCarthy, MD, Study Chair — Embera NeuroTherapeutics, Inc.
Locations (4):
- United States (4):
  - Pacific Treatment and Research Center, Department of Psychiatry, University of California, San Diego, School of Medicine, San Diego, California
  - Segal Trials, Miami, Florida
  - U PENN- Perelman School of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Every three months, the NIDA DSMB will convene to review the overall safety data, as well as data on safety summarized by treatment condition. As per NIH guidelines, the objective of these reviews will be to determine whether continued conduct of the trial poses any undue risk for participants. Blinded data tables, figures and/or listings will be provided to the Data Safety Monitoring Board (DSMB).
Supporting Information: Study Protocol, CSR
Time Frame: Every three months- blinded results
Access Criteria: A DSMB report is prepared an submitted via NIDA

REFERENCES:
- [Background] Kablinger AS, Lindner MA, Casso S, Hefti F, DeMuth G, Fox BS, McNair LA, McCarthy BG, Goeders NE. Effects of the combination of metyrapone and oxazepam on cocaine craving and cocaine taking: a double-blind, randomized, placebo-controlled pilot study. J Psychopharmacol. 2012 Jul;26(7):973-81. doi: 10.1177/0269881111430745. Epub 2012 Jan 11. PMID 22236504